CLINICAL TRIAL: NCT05050487
Title: Pericapsular Nerve Group Block Versus Lumber Erector Spinae Plane Block for Pain Management After Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdeltwab Younis Tamam, assisstant lecturer of anesthesia and intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: T1991
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Post Operative Pain, Chronic
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomized controlled trail
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): patient will recieve pericapsular nerve group block
  Interventions: Procedure: PENG block
- treatement (Experimental): patient will receive lumbar erector spinae plane block
  Interventions: Procedure: lumbar erector spinae plane block

INTERVENTIONS:
Procedure: PENG block — The PENG block is performed under US guid¬ance, . The pa¬tient is placed in the supine position a curvilinear low-fre¬quency ultrasound probe (2-5 MHz) is initially placed in a transverse plane over the AIIS and then aligned with the pubic ramus by rotating the probe approximately 30-45 degrees . .
  The needle, usually a 22-G80-mm echogenic device, is inserted from lateral to medial with an in-plane approach to place the tip in the plane between the psoas tendon anteriorly and the pu¬bic ramus posteriorly .
  After needle insertion and following negative aspiration, the local anesthetic is injected . The volume used of 20 ml of(L-bupivacaine; concentration 0,25% ) . This fascial plane appeared to continue in the hip pericapsular plane.
  Other Names: pericapsular nerve group block
  Arms: treatment
Procedure: lumbar erector spinae plane block — The lumbar erector spinae block is performed under US guid¬ance, after adequate skin disinfection The patient is placed in the lateral decubitus position according to the selected site of surgical intervention.
  The 4th lumbar vertebral level will determined The convex USG transducer was placed at the mid-vertebral line in the sagittal plane. The transducer was shifted from the midline, 3.5-4 cm laterally to the side of the surgery to visualize the erector spinae muscle and transverse process . 0.5-1 ml of the prepared LA solution (20 ml bupivacaine 0.25%). All LA was administered to this location between the transverse process and the erector spinae muscle.
  Other Names: ESPB
  Arms: treatement

SUMMARY:
Pain is a major problem that has to be dealt with in case of hip fracture, as it presents an obstacle for examination, positioning for receiving neuroaxial anesthesia and postoperative mobility and physiotherapy. With the introduction of ultrasound in regional anesthesia and peripheral nerve blocks, regional analgesia float to the surface as a substitute for opioids with less side effects Lumbar erector spinae plane block has emerged as a reliable analgesic option for primary total hip arthroplasty (THA). In 2018, a new block was described, termed pericapsular nerve group block or PENG block, that selectively targets the articular branches of the femoral and obturator nerves while sparing their motor components

DETAILED DESCRIPTION:
Pain is a major problem that has to be dealt with in case of hip fracture, as it presents an obstacle for examination, positioning for receiving neuroaxial anesthesia and postoperative mobility and physiotherapy. With the introduction of ultrasound in regional anesthesia and peripheral nerve blocks, regional analgesia float to the surface as a substitute for opioids with less side effects Lumbar erector spinae plane block has emerged as a reliable analgesic option for primary total hip arthroplasty (THA). In 2018, a new block was described, termed pericapsular nerve group block or PENG block, that selectively targets the articular branches of the femoral and obturator nerves while sparing their motor components The pericapsular nerve group (PENG) block is an ultrasound-guided approach first de-scribed by Giron-Arango et al. for the blockade of the articular branches of the femoral (FN), obturator (ON) and accessory obturator (AON) nerve that provide sensory innervation to the an¬terior hip capsule. It has been developed as an alternative regional anesthesia technique for the management of acute pain after hip fractures, but its applications are expanding.

Currently, the PENG block has been used to control and reduce pain in hip-related procedures.

There are reports of PENG blocks used as surgical anesthetic techniques for hip arthroplasty (in combination with local anesthetic and intravenous analgesics) or hip arthroscopy (in combination with lateral femoral cutaneous nerve [LFCN] block). There is a report of a PENG block used as analgesic technique for sickle cell disease vaso-occlusive crisis and a PENG radiofrequency ablation for osteoarthritis analgesia. There are also reports about the use of a PENG block for non-hip related interventions, such as leg vein ligation and stripping, medial thigh surgery, prevention of adductor muscle spasm during transurethral resection of bladder and below-knee amputation in association with popliteal sciatic nerve block.These latter cases further extended the application of the PENG block beyond the hip-related area.

So far, most of the reports describe preoperative or postoperative single-shot blocks, while there are only few case reports of continuous PENG blocks.

Due to the novelty of this technique, there are still ongoing debates about the best injection point as well as the best anesthetic concentration and the total volume to be injected.

Defined in the last decade, erector spinae plane block (ESPB) is one of the more frequently used interfacial plans, and it has been the most discussed block among the recently defined techniques. Lumbar ESPB administered at lumbar levels is relatively novel and is a new horizon for regional anesthesia and pain practice.(14)

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade 1&2 &3
2. Adult patients (Age >18 yrs)
3. Eligible patients were aged 18 years or older, were admitted for hip arthroplasty (THA or HA) for femoral neck fracture, and had undergone a preoperative RA technique (PENG block or lumbar erector spinae plane block)

Exclusion Criteria:

1. Patients with chronic pain before surgery (taking opioids)
2. Patients with multiple trauma
3. Patients who could not assess pain reliably (dementia)
4. Patients who in anticoagulation
5. Patient refused
6. Infection at the side of injection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hour
  the time passed from block to the patient's first analgesic request in hours